CLINICAL TRIAL: NCT06369103
Title: Comparison of the Sedative Effects of Dexmedetomidine and Propofol During Peribulbar Anaesthesia in Patients Undergoing Vitrectomy Surgery: A Prospective Randomized Clinical Trial
Brief Title: The Sedative Effects of Dexmedetomidine VS Propofol During Peribulbar Anesthesia in Patients Undergoing Vitrectomy Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Dina Mahmoud Fakhry, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/03032024/Fakhry
Record Dates: First submitted 2024-04-08; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Patient; Satisfaction
Keywords: Sedative Effects; Dexmedetomidine; Propofol; Vitrectomy
MeSH Terms: conditions — Personal Satisfaction | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Active Comparator): Patients will receive dexmedetomidine at a dose of 0.5-1.0 mcg/kg over 5-10 minutes, then a maintenance infusion rate of 0.2-0.5 mcg/kg/min when the bispectral index (BIS) value is between 70 and 80.
  Interventions: Drug: Dexmedetomidine
- Propofol Group (Active Comparator): Patients will receive propofol at a dose of 0.25-0.5 mg/kg over 5-10 minutes, then a maintenance Infusion rate of 0.5-2 mg/kg/hr when the bispectral index (BIS) value is between 70 and 80.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive dexmedetomidine at a dose of 0.5-1.0 mcg/kg over 5-10 minutes, then a maintenance infusion rate of 0.2-0.5 mcg/kg/min when the bispectral index (BIS) value is between 70 and 80.
  Arms: Dexmedetomidine Group
Drug: Propofol — Patients will receive propofol at a dose of 0.25-0.5 mg/kg over 5-10 minutes, then a maintenance Infusion rate of 0.5-2 mg/kg/hr when the bispectral index (BIS) value is between 70 and 80.
  Arms: Propofol Group

SUMMARY:
The aim of the work to compare the Sedative Effects of Dexmedetomidine and Propofol during peribulbar anesthesia in patients undergoing vitrectomy surgery on hemodynamic, respiratory parameters, recovery profile, analgesic effects, post-operative cognitive function, patients satisfaction and adverse events.

DETAILED DESCRIPTION:
In ocular surgery, local anesthesia or regional anesthesia is generally preferred over general anesthesia because of quicker patient rehabilitation and the avoidance of possible complications from general anesthesia. However, even with these anesthesia techniques, pain, fear and anxiety are major predictors of lower patient satisfaction.

Vitrectomy surgery is one of the most common outpatient ophthalmic surgeries. It can be performed with peribulbar anesthesia and intravenous (IV) sedation support, allowing the procedure to be completed in most patients without the need for general anesthesia. Vitrectomy surgery is a painful and lengthy procedure; therefore, sedation is applied to reduce patient agitation, ensuring both surgical comfort and hemodynamic stability. However, various complications can arise during the perioperative period depending on the sedation agent used.

Intravenous sedation is frequently used during ophthalmic regional anesthesia. There is no 'ideal' drug for sedation or analgesia. Various drugs either alone or in combination have been used with different methods of administration. The preferred sedative agent for ophthalmic surgeries performed under local anesthesia should have rapid onset but a short duration of action to ensure rapid recovery. It should be non-accumulating, non-toxic and have a favorable therapeutic index with minimal side effects. Unfortunately no drug is presently available that fulfils all these criteria. The available sedative drugs are benzodiazepines, intravenous anaesthetic induction agents (e.g. propofol), opiates and α-adrenoreceptor agonists such as dexmedetomidine or clonidine.

Among anesthetic agents, Dexmedetomidine is a strong selective α2-adrenergic agonist with sympatholytic, anxiolytic, analgesic and dose-dependent sedative/hypnotic properties, without causing respiratory depression.

Moreover, the use of dexmedetomidine reduces anesthetic and opioid requirements and also psychomotor function to be reserved.

Dexmedetomidine is the preferred agent for sedation in retinal surgery because of its ability to maintain hemodynamic and respiratory stability.

On the other hand, Propofol is an important intravenous anesthetic agent that has been extensively used as a sedative agent for ophthalmic procedures due to its favorable pharmacokinetic properties. Propofol has short duration of action, no cumulative effect, unique recovery profile as well as rapid emergence and anti-emetic properties. Respiratory depression and reduced blood pressure are major side effects of propofol. However, it has been suggested that propofol may still be safely administered if given at a lower dose. Other side effects of propofol include pain on injection, increased oculocardiac reflex, anaphylaxis and patient movement.

Despite many benefits, propofol sedation has been involved in producing the photic sneezing reflex induced by periocular injections of anesthetics.

Unexpected or sudden sneezing during injection can be a dangerous side effect in periocular injection, in which abrupt head movement may cause globe injury.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-70 years.
* Expected time of surgery less than 2 hours

Exclusion Criteria:

* patients with an initial mini mental state examination (MMSE) score less than 23
* Patients refusing LA
* Clotting abnormalities
* Impaired mental status
* Allergy to any of the study medications
* Also, patients were excluded if they had severe cardiac disease, chronic obstructive lung disease, a history of sleep apnea and those who received general anesthesia.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 6 hours after the end of surgery.
  Patient satisfaction will be also assessed using 7-point Likert-like verbal rating scale. One means extremely dissatisfied and seven means extremely satisfied.

SECONDARY OUTCOMES:
Visual analogue scale | 6 hours after the end of surgery
  The degree of pain was assessed by using a 10-cm visual analog scale (VAS) for pain where: 0=no pain and 10=intolerable pain

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Fakhry, MD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni Suef University Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt